CLINICAL TRIAL: NCT04169789
Title: Prevention of Early Postmenopausal Bone Loss With Lactobacillus Reuteri - A Randomized, Placebo-Controlled, Single Centre Clinical Trial
Brief Title: Prevention of Early Postmenopausal Bone Loss With Lactobacillus Reuteri
Acronym: ELBOWII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Mattias Lorentzon, Professor, Chief Physician, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELBOWII
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L. reuteri Low Dose (Active Comparator): Capsules of freeze-dried L. reuteri 6475 of 5x10E8 colony-forming units (CFU) mixed with maltodextrin powder and 200 IU of cholecalciferol, taken twice daily for 24 months, yielding a total dose of either 1x10E9 L.reuteri CFU and 400 IU of cholecalciferol per day.
  Interventions: Dietary Supplement: Lactobacillus reuteri ATCC PTA 6475 (L. reuteri 6475)
- L. reuteri High Dose (Active Comparator): Capsules of freeze-dried L. reuteri 6475 of 5x10E9 colony-forming units (CFU) mixed with maltodextrin powder and 200 IU of cholecalciferol, taken twice daily for 24 months, yielding a total daily dose of 1x10E10 L.reuteri CFU and 400 IU of cholecalciferol per day.
  Interventions: Dietary Supplement: Lactobacillus reuteri ATCC PTA 6475 (L. reuteri 6475)
- Placebo (Placebo Comparator): Placebo product identical to the active product (L. reuteri) in taste and appearance but without the active component, orally twice daily, for 24 months.The placebo product contains 200 IU cholecalciferol per dose, yielding a total dose of cholecalciferol of 400 IU per day.
  Interventions: Dietary Supplement: Lactobacillus reuteri ATCC PTA 6475 (L. reuteri 6475)

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri ATCC PTA 6475 (L. reuteri 6475) — L.reuteri high or low dose with cholecalciferol compared to cholecalciferol only.

SUMMARY:
This study evaluates the effect of two different doses of Lactobacillus reuteri ATCC PTA 6475 (L.reuteri 6475) on bone loss in early postmenopausal women. One third of the participants will be randomised to the lower dose, one third to the higher dose and one third to placebo.

DETAILED DESCRIPTION:
We have previously shown that daily supplementation of the probiotic Lactobacillus reuteri ATCC PTA 6475 (10E10 colony-forming units (CFU)) was able to reduce bone loss over 12 months in 76-year-old women compared to placebo.

It is not known if the probiotic is effective over longer time periods or if the effect is dose-dependent. The aim of this study is to investigate if two different doses of Lactobacillus reuteri ATCC PTA 6475 (total daily dose of either 1x10E9 or 1x10E10 CFU/day) can prevent or reduce bone loss, compared to placebo, in early (1-4 years since last menses) postmenopausal women over 24 months. All women will receive 400 IU of vitamin D (cholecalciferol) per day. Changes in bone mineral density, bone geometry and microstructure will be measured using dual x-ray absorptiometry and high resolution peripheral computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, 45 years or older, within 1-4 years from their last menses.
* Vitamin D levels above 25 nmol/L.
* Signed informed consent.
* Stated availability throughout the entire study period.
* Ability to understand study instructions and willingness to adhere to the protocol.

Exclusion Criteria:

* Bone mineral density of < -2.5 combined with a fracture risk assessment tool (FRAX) score of 20% or higher for major osteoporotic fracture.
* Severe osteoporosis, defined as bone mineral density of < -3.0 in either the total hip, femur neck or lumbar spine L1-L4.
* Vertebral fracture (grade II or III) diagnosed using lateral spine imaging with DXA.
* Untreated hyperthyroidism or hyperthyroidism within the last 5 years.
* Known untreated hyperparathyroidism.
* Rheumatoid arthritis.
* Diagnosed with disease causing secondary osteoporosis, including chronic obstructive pulmonary disease, inflammatory bowel disease, celiac disease, or diabetes mellitus.
* Recently diagnosed malignancy (within the last 5 years).
* Oral corticosteroid use.
* Previous (within the last 5 years) use of antiresorptive therapy, including systemic hormone therapy (estrogen), bisphosphonates, strontium ranelate or denosumab.
* Systemic skeletal disease (including e.g. Paget's disease and osteogenesis imperfecta).
* Any systemic disease that could affect bone loss, as judged by the investigator.
* Use of teriparatide (current or during the last 3 years).
* Participation in other clinical trials.
* Current antibiotics treatment or within the last 2 months prior to inclusion.
* Current and within the past 2 months use of probiotic supplement
* Vitamin D deficiency (25-OH vitamin D<25 nmol/l)
* Hypo- or hypercalcemia.
* Osteosynthesis materials in both lower legs (tibia).

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Total tibia volumetric bone mineral density | 24 months
  Measured using high resolution peripheral computed tomography (HRpQCT), relative change 0-24 months

SECONDARY OUTCOMES:
Areal bone mineral density (aBMD) at the lumbar spine | 24 months
  Measured using dual x-ray absorptiometry (DXA), relative change 0-24 months and 0-12 months
Areal BMD of the total hip (DXA) | 0-24 months and 0-12 months
  Measured using DXA, relative change 0-24 months and 0-12 months
Tibia trabecular bone volume fraction | 0-24 months and 0-12 months
  Measured using HRpQCT, relative change 0-24 months and 0-12 months
Tibia cortical area | 0-24 months and 0-12 months
  Measured using HRpQCT, relative change 0-24 months and 0-12 months
Tibia cortical volumetric BMD | 0-24 months and 0-12 months
  Measured using HRpQCT, relative change 0-24 months and 0-12 months
Total tibia volumetric bone mineral density | 12 months
  Measured using HRpQCT, relative change 0-12 months
Blood bone formation marker procollagen type 1N propeptide (P1NP) | 0-24 months and 0-12 months
  Relative change 0-24 months and 0-12 months
Blood bone resorption marker C-terminal cross-linking telopeptide of type I collagen (CTX) | 0-24 months and 0-12 months
  Relative change 0-24 months and 0-12 months
Fecal calprotectin | 0-24 months and 0-12 months
  Relative change 0-24 months and 0-12 months
Fecal lipocalin-2 | 0-24 months and 0-12 months
  Relative change 0-24 months and 0-12 months
Serum butyrate concentration | 0-24 months and 0-12 months
  Relative change 0-24 months and 0-12 months
Serum Wnt10b concentration | 0-24 months and 0-12 months
  Relative change 0-24 months and 0-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Lorentzon, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Geriatric Medicine, Sahlgrenska University Hospital, Mölndal, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsson AG, Sundh D, Backhed F, Lorentzon M. Lactobacillus reuteri reduces bone loss in older women with low bone mineral density: a randomized, placebo-controlled, double-blind, clinical trial. J Intern Med. 2018 Sep;284(3):307-317. doi: 10.1111/joim.12805. Epub 2018 Jul 22. PMID 29926979
- [Derived] Gregori G, Pivodic A, Magnusson P, Johansson L, Hjertonsson U, Brattemark E, Lorentzon M. Limosilactobacillus reuteri 6475 and Prevention of Early Postmenopausal Bone Loss: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2415455. doi: 10.1001/jamanetworkopen.2024.15455. PMID 38865129